CLINICAL TRIAL: NCT01082393
Title: Vitiligo and the Koebner Phenomenon (Model of Vitiligo Induction and Therapy: a Clinical and Immunological Analysis)
Acronym: Koebner
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/599
Record Dates: First submitted 2010-02-26; First posted 2010-03-08 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Vitiligo
Keywords: vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- topical tacrolimus (Active Comparator)
  Interventions: Drug: topical tacrolimus treatment
- topical pimecrolimus (Active Comparator)
  Interventions: Drug: topical pimecrolimus treatment
- local steroids (Active Comparator)
  Interventions: Drug: local mometasone furoate treatment
- cold cream (Placebo Comparator)
  Interventions: Drug: cold cream

INTERVENTIONS:
Drug: topical tacrolimus treatment — 4 applications (day 1,day 3, day 6 and day10)
  Arms: topical tacrolimus
Drug: topical pimecrolimus treatment — 4 applications (day 1, day 3, day 6 and day 10)
  Arms: topical pimecrolimus
Drug: local mometasone furoate treatment — 4 applications (day 1, day 3, day 6 and day 10)
  Arms: local steroids
Drug: cold cream — 4 applications (day 1, day 3, day 6 and day 10)
  Arms: cold cream

SUMMARY:
We will investigate the process of vitiligo induction and the influence of different commonly used cream treatments on this process. Studies comparing different treatments for vitiligo in the induction stage of the disease are still missing. The study hypothesis = cream treatment can stop actively spreading vitiligo lesions during the early induction stage of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female,
* Age 18-70 years,
* Extensive vitiligo (> 50% body surface area),
* Patients asking for depigmenting therapy,
* Not pregnant.

Exclusion Criteria:

* Children,
* Non extensive vitiligo (< 50% boy surface area),
* Patients not asking for depigmenting therapies,
* Pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02-16 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
percentage of skin pigmentation in the treated area | after 1 day, 10 days, 30 days and 60 days
  digital image analysis system for surface measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nanny Van Geel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be